CLINICAL TRIAL: NCT03015064
Title: Post-Myocardial Infarction Patients in Santa Catarina, Brazil: a Prospective Cohort Study - Catarina Heart Study
Brief Title: Post-Myocardial Infarction Patients in Santa Catarina, Brazil - Catarina Heart Study
Acronym: Catarina
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto de Cardiologia de Santa Catarina (Other)
Responsible Party: Principal Investigator, Daniel Medeiros Moreira, Clinical vice-director, Instituto de Cardiologia de Santa Catarina
Other Study IDs: CAAE: 55450816.0.1001.0113
Record Dates: First submitted 2016-12-30; First posted 2017-01-09 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial Infarction: Patients with first myocardial Infarction
  Interventions: Other: Myocardial Infarction

INTERVENTIONS:
Other: Myocardial Infarction — Observational study of myocardial Infarction patients

SUMMARY:
Prospective cohort evaluating patients in the State of Santa Catarina (Brazil) with the diagnosis of the first acute myocardial infarction from July 2016 until December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Presence of precordial pain suggestive of acute myocardial infarction associated with electrocardiogram with new ST segment elevation in two contiguous leads with limits: ≥0.1 mv in all leads other than leads V2-V3 where the following limits apply : ≥0.2 mv in Men ≥40 years; ≥0.25 mV in men <40 years, or ≥ 0.15 mV in women or presence of precordial pain suggestive of acute myocardial infarction associated with elevation of troponin I or CK-MB above the 99th percentile of the upper reference limit

Exclusion Criteria:

* Previous acute myocardial infarction;
* Disagreement with the Terms of Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attended at the Santa Catarina Institute of Cardiology and other hospitals in the State of Santa Catarina with the diagnosis of the first acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 1426 (Estimated)
Dates: Start 2016-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MACE in 1 year | Major cardiovascular events - MACE (cardiovascular death, nonfatal infarction, unstable angina or stroke) in 1 year
MACE in 30 days | Major cardiovascular events - MACE (cardiovascular death, nonfatal infarction, unstable angina or stroke) in 30 days
Death in 1 year | Death incidence in 1 year
Death in 30 days | Death incidence in 30 days
Restenosis in 1 year | Restenosis incidence in 1 year
Restenosis in 30 days | Restenosis incidence in 30 days
Intrastent thrombosis in 1 year | Intrastent thrombosis incidence in 30 days
Intrastent thrombosis in 30 days | Intrastent thrombosis incidence in 30 days
Cardiovascular death in 1 year | Cardiovascular death incidence in 1 year
Cardiovascular death in 30 days | Cardiovascular death incidence in 30 days
Nonfatal infarction in 1 year | Nonfatal infarction incidence in 1 year
Nonfatal infarction in 30 days | Nonfatal infarction incidence in 30 days
Unstable angina in 1 year | Unstable angina incidence in 1 year
Unstable angina in 30 days | Unstable angina incidence in 30 days
Stroke in 1 year | Stroke incidence in 1 year
Stroke in 30 days | Stroke incidence in 30 days

SECONDARY OUTCOMES:
Epidemiological profile | Epidemiological profile of hospitalized patients with infarction in Santa Catarina at the admission
Fish consumption | Fish consumption at admission
  Fish consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Red meat consumption | Red meat consumption at admission
  Read meat consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Chocolate consumption | Chocolate consumption at admission
  Red meat consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Caffeine consumption | Caffeine consumption at admission
  Caffeine consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Alcoholic beverages consumption | Alcoholic beverages consumption at admission
  Alcoholic beverages consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Illegal drugs consumption | Illegal drugs consumption at admission
  Illegal drugs consumption at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Cognitive level | Cognitive level at admission
  Cognitive level (evaluated with Mini-Mental State Examination) at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction syndromes and infarction
Religiosity | Religiosity at admission
  Religiosity (evaluated with Duke University Religion Index) at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Pre-infarct physical activity | Pre-infarct physical activity at admission
  Pre-infarct (evaluated with Baecke Questionnaire) physical activity at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Depression | Depression at admission
  Depression (evaluated with PHQ-9: Patient Health Questionnaire-9) at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Syntax score | Syntax score at admission
  Syntax score at admission and its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
TIMI frame count | TIMI frame count in patients with primary angioplasty at admission
  TIMI frame count in patients with primary angioplasty at admission its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Ventricular function post-infarction | Ventricular function post-infarction (evaluated within 72 hours of admission)
  Ventricular function (ventricular ejection fraction), its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction
Hospitalization in 1 year | Hospitalization incidence in 1 year
Hospitalization in 30 days | Hospitalization incidence in 30 days
Bleeding in 1 year | Bleeding incidence in 1 year
Bleeding in 30 days | Bleeding incidence in 30 days
Hematocrit and hemoglobin | Hematocrit and hemoglobin at the admission
Hematocrit and hemoglobin in 72 hours | Hematocrit and hemoglobin in 72 hours
Red Cell Distribution Width (RDW) | Red Cell Distribution Width (RDW) at admission
Red Cell Distribution Width (RDW) | Red Cell Distribution Width (RDW) in 72 hours
Leukocytes | Leukocytes at admission
Leukocytes | Leukocytes in 72 hours
Creatinine | Creatinine at admission
Creatinine | Creatinine in 72 hours
Troponin levels | Troponin levels at admission
Troponin levels | Troponin levels in 72 hours
Cholesterol levels | Cholesterol levels at admission
Cholesterol levels | Cholesterol levels in 72 hours
C-reactive protein | C-reactive protein at admission
C-reactive protein | C-reactive protein in 72 hours
CHA2DS2-VASc Score | CHA2DS2-VASc Score at admission
  CHA2DS2-VASc Score, its correlation with other evaluated parameters and its association with death, hospitalization, stroke, acute coronary syndromes and infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia de Santa Catarina, São José, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No